CLINICAL TRIAL: NCT03023293
Title: Effects and Mechanisms of n-3 Polyunsaturated Fatty Acids and Irisin on the Incidence of Abnormal Glucose Metabolism After Gestational Diabetes Mellitus
Brief Title: Effects and Mechanisms of n-3 PUFAs and Irisin on Abnormal Glucose Metabolism After GDM.
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Li Cai, Principal Investigator, Sun Yat-sen University
Other Study IDs: LCai
Record Dates: First submitted 2017-01-13; First posted 2017-01-18 (Estimated); Last update posted 2019-01-11 (Actual); Status verified 2019-01

CONDITIONS: Gestational Diabetes Mellitus
Keywords: n-3 polyunsaturated fatty acids; irisin
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — the status of n-3 polyunsaturated fatty acids and irisin in plasma/serum/eryhrocyte membrane.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- gestational diabetes mellitus: The investigators plan to establish a prospective GDM cohort and collect n-3 PUFAs consumption and irisin information at 24-28 weeks'gestation, 42 days postpartum, 1 year postpartum and 2 years postpartum, respectively.
  Interventions: Other: n-3 PUFAs consumption and irisin

INTERVENTIONS:
Other: n-3 PUFAs consumption and irisin — The investigators plan to collect n-3 PUFAs and irisin information at 24-28 weeks' gestation, 42 days postpartum, 1 year postpartum and 2 years postpartum

SUMMARY:
The purpose of this study is to clarify the relationship between n-3 PUFA and irisin in regulating the glucose metabolism in GDM patients.

DETAILED DESCRIPTION:
Gestational diabetes mellitus (GDM) is an important risk factor for type 2 diabetes in women. Studies have shown that n-3 polyunsaturated fatty acids (n-3 PUFA) are associated with improving insulin resistance and prevent type 2 diabetes in the general population; a newly discovered myokine, irisin, is associated with reduced insulin resistance and plays an important role in human glucose metabolism; and results from cell studies suggested that n-3 PUFA might increase the expression of irisin. Therefore, the investigators hypothesize that n-3 PUFA could improve glucose metabolism via the IRS-1/PI3K/AKT insulin signaling pathway by increasing expression of irisin and thus improving postpartum glucose metabolism in women with GDM. In order to test this hypothesis, the investigators plan to establish a prospective GDM cohort and collect related information at 24-28 weeks' gestation, 42 days postpartum, 1 year postpartum and 2 years postpartum, respectively. Then the following would be tested: the changes of n-3 PUFA and irisin during pregnancy and after delivery, and their association with postpartum abnormal glucose metabolism; and the correlation of n-3 PUFA and irisin. Furthermore, using a cell model of insulin resistance the investigators would examine the dose-response and time-response relationships between n-3 PUFA and irisin, and next explore the role of irisin in n-3 PUFA regulation of IRS-1/PI3K/AKT insulin signaling pathway. This study would help to clarify the relationship between n-3 PUFA and irisin in regulating the glucose metabolism, and might provide scientific evidence for the prevention of type 2 diabetes after GDM.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women with gestational diabetes mellitus were screened by The Guidelines for diagnosis and treatment of gestational diabetes mellitus in China in 2014.

Exclusion Criteria:

* age < 20 years or ≥ 45 years;
* women with diabetes, cardiovascular disease, thyroid disease, blood disease and polycystic ovary syndrome before pregnancy;
* multiple pregnancy and assisted reproductive technology pregnancy;
* women with severe postpartum endocrine disorders and diseases, such as pancreatitis, hyperthyroidism, nephritis;
* infection during pregnancy.

Ages: 20 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: pregnant women with gestational diabetes mellitus
Sampling Method: Probability Sample
Enrollment: 1285 (Estimated)
Dates: Start 2017-03-10 (Actual); Primary Completion 2019-04-05 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
postpartum glucose metabolism | during 2 years postpartum
  We will measure the glucose metabolism by OGTT.

CONTACTS AND LOCATIONS:
Overall Officials: Li Cai, Principal Investigator — Sun Yat-sen University
Locations (1):
- Weijia, Wu, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Villegas R, Xiang YB, Elasy T, Li HL, Yang G, Cai H, Ye F, Gao YT, Shyr Y, Zheng W, Shu XO. Fish, shellfish, and long-chain n-3 fatty acid consumption and risk of incident type 2 diabetes in middle-aged Chinese men and women. Am J Clin Nutr. 2011 Aug;94(2):543-51. doi: 10.3945/ajcn.111.013193. Epub 2011 Jun 15. PMID 21677058
- [Background] Nanri A, Mizoue T, Noda M, Takahashi Y, Matsushita Y, Poudel-Tandukar K, Kato M, Oba S, Inoue M, Tsugane S; Japan Public Health Center-based Prospective Study Group. Fish intake and type 2 diabetes in Japanese men and women: the Japan Public Health Center-based Prospective Study. Am J Clin Nutr. 2011 Sep;94(3):884-91. doi: 10.3945/ajcn.111.012252. Epub 2011 Jul 20. PMID 21775559
- [Background] Brostow DP, Odegaard AO, Koh WP, Duval S, Gross MD, Yuan JM, Pereira MA. Omega-3 fatty acids and incident type 2 diabetes: the Singapore Chinese Health Study. Am J Clin Nutr. 2011 Aug;94(2):520-6. doi: 10.3945/ajcn.110.009357. Epub 2011 May 18. PMID 21593505
- [Background] Zhao L, Li J, Li ZL, Yang J, Li ML, Wang GL. Circulating irisin is lower in gestational diabetes mellitus. Endocr J. 2015;62(10):921-6. doi: 10.1507/endocrj.EJ15-0230. Epub 2015 Jul 29. PMID 26228794
- [Background] Kuzmicki M, Telejko B, Lipinska D, Pliszka J, Szamatowicz M, Wilk J, Zbucka-Kretowska M, Laudanski P, Kretowski A, Gorska M, Szamatowicz J. Serum irisin concentration in women with gestational diabetes. Gynecol Endocrinol. 2014 Sep;30(9):636-9. doi: 10.3109/09513590.2014.920006. Epub 2014 May 22. PMID 24850254
- [Background] Vaughan RA, Garcia-Smith R, Bisoffi M, Conn CA, Trujillo KA. Conjugated linoleic acid or omega 3 fatty acids increase mitochondrial biosynthesis and metabolism in skeletal muscle cells. Lipids Health Dis. 2012 Oct 30;11:142. doi: 10.1186/1476-511X-11-142. PMID 23107305
- [Derived] Tang N, He Y, Karatela S, Zhong J, Zeng X, Lu Q, Zhao F, Cai L. Association between erythrocyte polyunsaturated fatty acids and gestational diabetes mellitus in Chinese pregnant women. Eur J Nutr. 2025 Feb 11;64(2):87. doi: 10.1007/s00394-025-03603-2. PMID 39932572